CLINICAL TRIAL: NCT03652727
Title: Appropriateness of Replacing Fluoroscopic Guidance by ECG Guidance in PICC Insertion, RCT
Brief Title: FX vs. ECG Guidance for PICC Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salah D. Qanadli (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor-Investigator, Salah D. Qanadli, Prof. MD PhD, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-00907
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Long Term Antibiotics; Chemotherapy; Total Parenteral Nutrition
Keywords: PICC; PIC Line; ECG
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECG-EM Guidance (Experimental): PICC insertion using electrocardiographic and electromagnetic guidance [Site~Rite® 8 Ultrasound System with integrated SHERLOCK 3CG™ Diamond Tip Confirmation System (TCS)]
  Interventions: Device: ECG-EM Guidance
- FX Guidance (Active Comparator): PICC insertion using fluoroscopic guidance
  Interventions: Device: FX Guidance

INTERVENTIONS:
Device: ECG-EM Guidance — ECG-EM method consists on a puncture of an arm vein, under the ultrasound control and local anesthesia. The length of the PICC is estimated prior to its insertion using morphological landmarks. The placement of the PICC is done using SHERLOCK 3CG™ Diamond Tip Confirmation System (TCS) [CE marked device, C. R. Bard, Inc.].
  At the end of procedure, a chest x-ray is performed to assess the PICC position
  Arms: ECG-EM Guidance
Device: FX Guidance — FX method consists on a puncture of an arm vein, under the ultrasound control and local anesthesia. Through the point of puncture, a long wire is then introduced and directed to the level of the target zone located in the superior vena cava under fluoroscopy control. The length of the guide inside the vessel is then measured to adjust the length of the PICC necessary for its optimal positioning.
  At the end of procedure, a chest x-ray is performed to assess the PICC position
  Arms: FX Guidance

SUMMARY:
The aim of this study is to compare two techniques of placing a peripherally inserted central venous catheter (PICC). The first technique, uses ECG based electromagnetic guidance (ECG-EM). The second (reference technique), is guided by X-ray (fluoroscopy).

DETAILED DESCRIPTION:
The method of placement under fluoroscopic control (FX) is considered as the reference technique. This is often criticized for disadvantages such as costs, logistical problems and relative ionizing radiation. Despite this, it is still advised by 75% of PICC providers.

Appeared about ten years ago, a per procedural guiding technique with intracavitary ECG tracking (ECG-EM) presents a better technical success (precision and specificity) than the blind technique, but there is still a lack in comparing this technique to the FX technique.

This prospective randomized controlled study is designed to compare the PICC insertion using ECG-EM guidance to fluoroscopic (FX) guidance in order to define whether a replacement of the FX technique by ECG-EM is appropriate in terms of the final catheter tip position of the PICC as well as length of the outgoing catheter at the entry point.

All included patients gave their written consent and the study is approved by EC.

Participation is open to all adults referred to the radiology department of the CHUV for insertion of a PICC (monocentric).

Recruited patients will be randomly assigned to one of the two arms (FX or ECG-EM).

For both procedures patient position and preparation (MSB, maximal sterile barrier) are standardized and are similar.

FX method consists on a puncture of an arm vein, under the ultrasound control and local anesthesia. Through the point of puncture, a long wire is then introduced and directed to the level of the target zone located in the superior vena cava under fluoroscopy control. The length of the guide inside the vessel is then measured to adjust the length of the PICC necessary for its optimal positioning.

For ECG-EM insertion technique, the vein puncture is done in similar conditions to the FX method. The length of the PICC is estimated prior to its insertion using morphological landmarks. The placement of the PICC is done using SHERLOCK 3CG™ Diamond Tip Confirmation System (TCS) (CE marked device; C. R. Bard, Inc.).

At the end of procedure, a chest x-ray is performed to assess the PICC position. Possible per-procedural complications are documented.

After intervention, the patient is transferred back to the ward or sent home in stable conditions.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Informed Consent Form)
* Adult > 18 years
* Referred to the interventional radiology department for PICC insertion

Exclusion Criteria:

* Pregnant women
* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Impairment of the heart rhythm changing the presentation of the P wave (atrial fibrillation, atrial flutter, severe tachycardia, pacemaker driven rhythm)
* Enrolled in conflicting research study
* Weight> 150 kg, technical limit for the fluoroscopy table
* Impossibility of obtaining informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Tip to CAJ (Cavo-atrial junction) | Up to 1 hour, after the procedure
  At the end of intervention tip position is measured on chest fluoroscopic X-ray.
  Absolute distance from tip to CAJ is measured on the image. This will reflect proportions of optimal tip positions depending on guidance technology.
  Rationale is that optimal position is mandatory for adequate functioning of PICC as malpositions may result on cardiac rhythm disorders, thrombosis or premature PICC occlusion.

SECONDARY OUTCOMES:
Length of the outgoing catheter | Up to 1 hour, after the procedure
  Length of the outgoing catheter at the entry point near the bend of the elbow. The rationale behind is that correct positioning guarantees optimal haemostasis and might prevent secondary displacement
Inter-observer and intra-observer variance | Through study completion, an average of 9 month
  The CAJ to catheter tip distance is based on subjective assessment by one investigator of the X-ray chest. Rationale behind is that in order to evaluate the impact of potential variation due to subjective interpretation interobserver and intraobserver variance will be quantified

CONTACTS AND LOCATIONS:
Overall Officials: Salah Dine Qanadli, Prof. MD PhD, Study Director — UNIL-CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gullo G, Colin A, Frossard P, Jouannic AM, Knebel JF, Qanadli SD. Appropriateness of Replacing Fluoroscopic Guidance With ECG-Electromagnetic Guidance for PICC Insertion: A Randomized Controlled Trial. AJR Am J Roentgenol. 2021 Apr;216(4):981-988. doi: 10.2214/AJR.20.23345. Epub 2021 Feb 17. PMID 33594912